CLINICAL TRIAL: NCT04337892
Title: Veracity Surgical: A Time/Motion and Quality of Care Study
Status: Completed | Type: Observational
Sponsor: Research Insight LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 200118
Record Dates: First submitted 2020-04-06; First posted 2020-04-08 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2020-04

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Standard of Care4 — The current standard of care for surgical planning for the participating investigator surgeon is to use Zeiss Veracity Surgical, so this same method will be used for the surgery actually performed on participating patients.

SUMMARY:
This study aims to compare the time required for surgical planning using these two methods and to explore whether differences in surgical accuracy can be identified in a small study of 40 patients.

DETAILED DESCRIPTION:
This study aims to compare the time commitment for surgical planning using these two methods and to explore whether differences in surgical accuracy can be identified in a small study of 40 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age with upcoming cataract surgery. At least 25% of enrolled eyes must be post-refractive, and 25% must require astigmatic planning (arcuate incision or toric IOL)
* Patients with otherwise healthy eyes, not exhibiting any significant ocular morbidity that would be expected to influence refractive outcome or interfere with postoperative refraction accuracy.

Exclusion Criteria:

* Patients with visually significant comorbidities (corneal, retina, optic nerve disease, not including prior refractive surgery) that could significantly affect their ability to have accurate preoperative biometry or postoperative refraction.
* Patients with surgical complications either during or after surgery (capsule tears, iris trauma, decentered IOL, cystoid macular edema, etc.) that would interfere with postoperative refraction.
* Patients with > grade 2 or greater posterior capsule opacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study aims to enroll 40 patients undergoing future cataract surgery.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Average number of minutes:seconds to plan surgery for a single eye | 1 day

SECONDARY OUTCOMES:
By each method the number of total data points where a human is required manually to transcribe data from one place to another. | 1 day

OTHER OUTCOMES:
Exploratory Endpoint: By each method the % of patients within 0.5 D of the intended postoperative manifest spherical equivalent refraction | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: John Hovanesian, MD, Study Director — Research Insight LLC
Locations (1):
- Harvard Eye Associates, Laguna Hills, California, United States

IPD SHARING:
Plan to Share IPD: No